CLINICAL TRIAL: NCT02228863
Title: Upper Extremity Rehabilitation Using Robot and Botulinum Toxin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2014-01-005
Record Dates: First submitted 2014-08-23; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Stroke; Spasticity
Keywords: Stroke; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Early Inmotion and Botox (Experimental): Concomitant use of Inmotion and botulinum toxin from the baseline
  Interventions: Other: Early Inmotion and Botox
- Botox, then Inmotion (Active Comparator): Inmotion training 4 weeks after botulinum toxin injection
  Interventions: Other: Botox, then Inmotion
- Inmotion, then Botox (Active Comparator): From the baseline Inmotion, then Botox injection at 4 weeks after baseline
  Interventions: Other: Inmotion, then Botox
- Late Inmotion and Botox (Active Comparator): No intervention, then Inmotion and Botox injection at 4 weeks from the baseline
  Interventions: Other: Late Inmotion and Botox

INTERVENTIONS:
Other: Early Inmotion and Botox — Concomitant use of Inmotion and Botox from the baseline
  Arms: Early Inmotion and Botox
Other: Botox, then Inmotion — At baseline Botox injection and 4 weeks after Inmotion
  Arms: Botox, then Inmotion
Other: Inmotion, then Botox — Inmotion from the baseline, then Botox injection at 4 weeks after baseline
  Arms: Inmotion, then Botox
Other: Late Inmotion and Botox — No intervention until 4 weeks from the baseline. Then Inmotion and Botox injection
  Arms: Late Inmotion and Botox

SUMMARY:
Concomitant use of botulinum toxin and robot would make better results regarding upper extremity function compared to robot, botulinum toxin, or no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Shoulder or Elbow flexor spasticity above or modified ashworth scale 1+
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* History of surgery of affected upper limb
* Fracture of affected upper limb
* Recent history of botulinum toxin injection within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Change of Fugl-Meyer Assessment | Fugl-Meyer Assessment change from baseline at 8 weeks

SECONDARY OUTCOMES:
Kinematic data | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
  Kinematic data from motion analysis (Vicon) Kinematic data from Inmotion
Spasticity of elbow and shoulder joint | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
  Modified Ashworth scale of elbow and shoulder joint Modified Tardieu scale of elbow and shoulder joint
Medical research council scale of elbow and shoulder joint strength | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
Painless range of motion of elbow and shoulder joint | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
numeric rating scale of pain of elbow and shoulder joint | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
Associated reaction rating scale | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
surface electromyography data from bilateral upper extremities | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
Behavioral activation system/behavioral inhition system scale | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
  In terms of motivation
Controlled Oral Word Association Test | baseline, 5ays of Inmotion, 20 days of Inmotion
  Controlled Oral Word Association Test during baseline, 5 days of Inmotion, 20 days of Inmotion.
  The test was done at rest and with Inmotion trial
Fugl-Meyer Assessment | Baseline, 4 weeks from baseline, 8 weeks from baseline, 12 weeks from baseline
Stroke impact scale | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
Beck's depression index | baseline, 4 weeks, 8 weeks, and 12 weeks from baseline
Satisfaction about the intervention | baseline, 4 weeks after baseline, 8 weeks after baseline, 12 weeks after baseline
Adverse event | From baseline to 12 weeks from the baseline
Digit span test | baseline, 5days after Inmotion, 20 days after Inmotion.
  Digit span test(forward, backward) during baseline, 5 days of Inmotion, 20 days of Inmotion.
  The test was done at rest and with Inmotion trial

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Shin JH, Park G, Kim H, Cho DY, Kwon S. Combined effects and timing of robotic training and botulinum toxin on upper limb spasticity and motor function: a single-blinded randomized controlled pilot study. J Neuroeng Rehabil. 2025 Mar 6;22(1):50. doi: 10.1186/s12984-025-01584-1. PMID 40050906
- See also: Site of the present study — http://nrc.go.kr